CLINICAL TRIAL: NCT02323672
Title: Salivary and Serum Levels of Chemerin and MMP-9 in Oral Precancer and Oral Squamous Cell Carcinoma.
Brief Title: Salivary and Serum Levels of Chemerin and MMP-9 in Oral Premalignant and Malignant Lesions
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of periodontology and Oral Medicine, faculty of oral and dental medicine, Cairo University
Other Study IDs: chemerin_MMP-9_Oral_cancer
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Precancerous Conditions; Oral Cancer
MeSH Terms: conditions — Precancerous Conditions; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and whole unstimulated saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- oral premalignant patients: 15 patients suffering from oral premalignant lesions as lichen planus, actinic keratosis, leukoplakia and erythroplakia.
- oral malignant patients: 15 patients suffering from oral malignant lesions
- control subjects: 15 individuals age, gender and periodontal status matched with oral premalignant and malignant patients and not suffering from any oral mucosal lesions or periodontal disease.

SUMMARY:
45 individuals were subdivided into 3 groups, 15 patients with oral premalignant lesions, 15 patients with oral malignant lesions and 15 control individuals. Levels of chemerin and MMP-9 were evaluated in serum and saliva of these subjects utilizing the ELISA technique.

DETAILED DESCRIPTION:
45 individuals were subdivided into 3 groups, 15 patients suffering from oral premalignant lesions, 15 patients suffering from oral malignant lesions and 15 individuals having age, gender and periodontal status matched with both patients groups acting as a control group. Serum and whole unstimulated saliva samples were collected from all the included groups in order to determine chemerin and MMP-9 in serum and saliva utilizing the ELISA technique.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral premalignant lesions.
* patients with oral malignant lesions.

Exclusion Criteria:

* any systemic disease other than oral premalignant or malignant lesions. smokers. pregnant females. periodontal diseases.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 45 individuals were subdivided into 3 groups, 15 patients suffering from oral squamous cell carcinoma lesions, 15 patients suffering from oral premalignant lesions (OPL) and 15 individuals having age, gender and periodontal status matched with both patients groups acting as a control group.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
salivary levels of chemerin in patients with oral premalignant and malignant lesions. | 1 day

SECONDARY OUTCOMES:
serum levels of chemerin in patients with oral premalignant and malignant lesions. | 1 day
serum levels of MMP-9 in patients with oral premalignant and malignant lesions. | morning visit
salivary levels of MMP-9 in patients with oral premalignant and malignant lesions. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ghallab, M.D., Principal Investigator — Associate Professor of periodontology and Oral Medicine faulty of oral and dental medicine Cairo Unv.

REFERENCES:
- [Background] Skrzeczynska-Moncznik J, Stefanska A, Zabel BA, Kapinska-Mrowiecka M, Butcher EC, Cichy J. Chemerin and the recruitment of NK cells to diseased skin. Acta Biochim Pol. 2009;56(2):355-60. Epub 2009 Jun 18. PMID 19543554
- [Background] Parolini S, Santoro A, Marcenaro E, Luini W, Massardi L, Facchetti F, Communi D, Parmentier M, Majorana A, Sironi M, Tabellini G, Moretta A, Sozzani S. The role of chemerin in the colocalization of NK and dendritic cell subsets into inflamed tissues. Blood. 2007 May 1;109(9):3625-32. doi: 10.1182/blood-2006-08-038844. Epub 2007 Jan 3. PMID 17202316
- [Background] Zhou XJ, Sugerman PB, Savage NW, Walsh LJ. Matrix metalloproteinases and their inhibitors in oral lichen planus. J Cutan Pathol. 2001 Feb;28(2):72-82. doi: 10.1034/j.1600-0560.2001.280203.x. PMID 11168755
- [Background] Nanda DP, Dutta K, Ganguly KK, Hajra S, Mandal SS, Biswas J, Sinha D. MMP-9 as a potential biomarker for carcinoma of oral cavity: a study in eastern India. Neoplasma. 2014;61(6):747-57. doi: 10.4149/neo_2014_091. PMID 25150320
- [Background] Wang N, Wang QJ, Feng YY, Shang W, Cai M. Overexpression of chemerin was associated with tumor angiogenesis and poor clinical outcome in squamous cell carcinoma of the oral tongue. Clin Oral Investig. 2014 Apr;18(3):997-1004. doi: 10.1007/s00784-013-1046-8. Epub 2013 Jul 19. PMID 23868294